CLINICAL TRIAL: NCT04683666
Title: Cardiovascular Risk Factors of Medical and Septic Complications After Laparoscopic Bariatric Surgery. A Prospective Cohort Study
Brief Title: Cardiovascular Risk Factors of Medical and Septic Complications After Laparoscopic Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: Hospital General Universitario Elche (Other)
Collaborators: Dr. Negrin University Hospital (Other)
Responsible Party: Principal Investigator, Jaime Ruiz-Tovar, MD, PhD, Clinical Professor, Hospital General Universitario Elche
Other Study IDs: CEIC13-2
Record Dates: First submitted 2020-12-21; First posted 2020-12-24 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Complication of Surgical Procedure
MeSH Terms: interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Bariatric surgery — Laparoscopic Roux-en-Y gastric bypass (LRYGB) or laparoscopic sleeve gastrectomy (LSG), as primary bariatric procedures, were performed. ^Postoperative complications were assessed.

SUMMARY:
A prospective, observational study of all morbidly obese patients undergoing laparoscopic Roux-en-Y gastric bypass (LRYGB) or laparoscopic sleeve gastrectomy (LSG) was performed. We evaluated preoperative comorbidities and cardiovascular risk factors, and the appearance of postoperative complications up to 90 days after surgery.

DETAILED DESCRIPTION:
This study aimed to identify potential cardiovascular risk factors for postoperative medical and septic complications after bariatric surgery.

A prospective, observational study of all morbidly obese patients undergoing laparoscopic Roux-en-Y gastric bypass (LRYGB) or laparoscopic sleeve gastrectomy (LSG) was performed. We evaluated preoperative comorbidities and cardiovascular risk factors, and the appearance of postoperative complications up to 90 days after surgery.

Evaluated cardiovascular risk factors include age, the presence of tobacco habit, preoperative diagnosis of T2D, hypertension, dyslipidemia, cardiopathies (including arrhythmias, ischemic cardiopathy or congestive cardiac failure), strokes, Charlson index and analytical parameters of the lipid (triglycerids, total cholesterol and the subfractions High Density Lipoproteins (HDL-cholesterol) and Low Density Lipoproteins (LDL-cholesterol) and glycemic profile (fasting glucose and glycated hemoglobin). Cardiovascular risk factors, such as the Framingham risk score, were analyzed.

Primary outcomes were the appearance of medical and septic postoperative complications. Medical complications include cardiovascular complications (new onset or impairment of acute heart infarction, arrhythmias, cardiac failure or stroke), respiratory complications (pneumonia or respiratory failure) and acute renal failure. Septic complications include, urinary tract infections, incisional or organ/space surgical site infection (SSI), pneumonia or bacteriemia of other origin.

ELIGIBILITY:
Inclusion Criteria:

* BMI >40 Kg/m2
* BMI >35 Kg/m2 associated with obesity-related comorbidities

Exclusion Criteria:

* ASA IV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients included were morbidly obese patients or patients with severe obesity associated with obesity-related comorbidities
Sampling Method: Non-Probability Sample
Enrollment: 177 (Actual)
Dates: Start 2013-03-15 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Medical complications | 90 days after surgery
  Medical complications include cardiovascular complications (new onset or impairment of acute heart infarction, arrhythmias, cardiac failure or stroke), respiratory complications (pneumonia or respiratory failure) and acute renal failure.
Septic complications | 90 days after surgery
  Septic complications include, urinary tract infections, incisional or organ/space surgical site infection (SSI), pneumonia or bacteriemia of other origin.

CONTACTS AND LOCATIONS:
Overall Officials: Asuncion Acosta, Study Director — Hospital Universitario Dr Negrin